CLINICAL TRIAL: NCT03780621
Title: Effects of an Adaptogenic Extract on Electrical Activity of Brain in Elderly Subjects With Cognitive Impairment: a Randomized, Double Blind, Placebo-controlled, Two Arms Cross-over Study.
Brief Title: Effects of an Adaptogenic Extract on Electrical Activity of the Brain in Elderly Subjects With Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-1004
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Cognitive Impairment, Mild
Keywords: Electroencephalography; Andrographis; Ashwagandha
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Andrographis and Withania (Experimental): Active ingredient: 550 mg of Andrographis paniculata (standardized to 40 mg andrographolides) and Withania somnifera (standardized to 10 mg withanolides) taken twice daily, once in the morning and once in the evening
  Interventions: Dietary Supplement: Andrographis and Withania
- Placebo (Placebo Comparator): 550 mg capsule visually identical to the active dietary supplement, containing brown sugar, microcrystalline cellulose, corn starch, and magnesium stearate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Andrographis and Withania — Combination of Andrographis paniculata and Withania somnifera
  Arms: Andrographis and Withania
Dietary Supplement: Placebo — Visually identical placebo capsule
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, two arm cross-over study to determine whether a specific combination of Andrographis paniculata and Withania somnifera can be regarded as a safe and effective treatment for cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers suffering from cognitive deficits.
* Questionnaire-DemTect. "DemTect" (for pre-selection of subjects) - score values 8-12 are regarded as conclusive.
* Age between 60 and 75 years (both included).
* Subjects should be right-handed.
* Subject must be capable of giving informed consent.
* Acceptance of written consent to participate in the study after instruction in written and oral form (informed consent).

Exclusion Criteria:

* Subjects with acute or chronic diseases that are relevant to the study and asked for by the study staff are excluded.
* Acute or chronic disease with an impact on the study, which becomes obvious by case history or clinical examination.
* Clinically relevant allergic symptoms.
* Detection of alcohol at the time of initial examination (day SC) or on study day A (positive alcohol test) or by case history.
* Consumption of clinically relevant medication during last 14 days before and during the active study period based on the notification of the subject or his case history.
* Consumption of medication with primarily central action (i.e. psychotropic drugs or centrally acting antihypertensive drugs). Known intolerance / hypersensitivity (allergy) to plant derived extracts or any of the ingredients of the investigational product (anamnestic).
* Presence of a rare, genetic disease such as fructose intolerance, glucose-galactose malabsorption or sucrose-isomaltase deficiency (anamnestic).
* Consumption of unusual quantities or misuse of coffee (more than 4 cups a day), tea (more than 4 cups a day).
* Detection of alcohol at the time of initial examination as well as on day A, B, C and D (alcohol test).
* Smoking in the study center on study days A, B, C and D.
* Result of the DemTect Questionnaire score <8 or >12.
* Participation in another clinical trial within the last 60 days.
* Bad compliance.
* Cancellation of informed consent.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change over time in neural electrical activity of the brain as measured by quantitative-topographic EEG for herbal treatment group versus placebo | Four weeks
  Responses of electric brain activity as spectral power in 17 different brain regions within 6 specially defined frequency ranges (delta, theta, alpha1, alpha2, beta1 and beta2) during the test of cognitive performance: d2-test for attention (d2-Test), memory test (ME-Test), concentration-performance-test with financial reward (CPT-Test).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Koch, MD, Principal Investigator — NeuroCode AG
Locations (1):
- Clinical Labors of NeuroCode AG, Wetzlar, Germany

IPD SHARING:
Plan to Share IPD: No